CLINICAL TRIAL: NCT00062777
Title: A Genome-Wide Scan for Quantitative Trait Loci of Hematocrit - A Framingham Study
Brief Title: The Framingham Study: Examining DNA Markers and Links to Diseases
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030219; 03-H-0219
Record Dates: First submitted 2003-06-13; First posted 2003-06-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-06-16

CONDITIONS: Vascular Diseases
Keywords: Genetics; Populations; CVD Risk; Gene Mapping; Epidemiology; Framingham Study; Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

SUMMARY:
Since 1948, residents of Framingham, Massachusetts, have participated in a program that collects blood samples and clinical data to provide a rare and valuable database for scientific research.

The purpose of this study is to support this national resource by aiding in its research capacity. Specifically, researchers in this study will (1) investigate heart, lung, and blood diseases; stroke; memory loss; joint disease; bone loss; deafness; cancer; blood vessel diseases and other health conditions, and (2) examine DNA and its relationship to risk of developing these disease and health conditions.

Approximately 330 families have participated in the Framingham Study. Participants will be required to undergo a four-hour exam and to take that exam every two years thereafter. During the exam, the Framingham investigators will (1) interview participants about medical status, health issues, and lifestyles; (2) perform a regular physical exam; (3) obtain blood and urine samples and administer a glucose-tolerance test; (4) supervise a brisk six-minute treadmill walk; (5) administer an ultrasound procedure; and (6) review and obtain copies of medical and hospital records. Participants will also be asked to complete a questionnaire at home regarding dietary and health habits.

DETAILED DESCRIPTION:
Many studies have shown that hematocrit (HCT) levels are associated with cerebrovascular disease, cardiovascular disease (CVD), peripheral vascular disease, as well as all-cause mortality. Twin studies have shown that HCT variation is largely determined by genetic factors with heritability estimated as 40% - 65%. So far, no linkage analysis in humans between HCT and DNA markers have been reported. The purpose of this protocol is to identify chromosome regions that contain quantitative trait loci (QTL) involved in controlling HCT levels. In the Framingham Study, a 10cM genome scan (about 400 markers) has been conducted in 330 families. HCT was measured in the original cohort and Framingham offspring. These data provide us the opportunity to undertake linkage analyses using variance component method to map quantitative trait loci (QTL) of HCT.

ELIGIBILITY:
* INCLUSION /EXCLUSION CRITERIA

The study population will include the members of the 330 Framingham Study families with genome scan.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2003-06-12; Study Completion 2011-06-16

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States